CLINICAL TRIAL: NCT02203864
Title: An Open-label, Multicenter, Controlled, Combined Parallel Group and Dose Escalation (0, 0.12, 1.2, 12.0 µg IL-2/10**8 Cells/24 Hours) Study, to Evaluate the Safety and Tolerability of an Allogeneic Tumor Vaccine BIWB 2 Containing Melanoma Cells Transfected With the Human IL-2 Gene in Patients With Advanced Malignant Melanoma
Brief Title: Dose Escalation Study to Evaluate Safety and Tolerability of an Allogeneic Tumor Vaccine BIWB 2 in Patients With Advanced Malignant Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1155.2
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

ARMS (2):
- BIBW2 with IL-2 secreting cell line (Experimental)
  Interventions: Biological: BIBW2 component B
- BIBW2 without IL-2 secreting cell line (Experimental)
  Interventions: Biological: BIBW2 component A

INTERVENTIONS:
Biological: BIBW2 component A — BIBW2 without IL-2 secreting cell line
  Arms: BIBW2 without IL-2 secreting cell line
Biological: BIBW2 component B — BIBW2 with IL-2 secreting cell line
  Arms: BIBW2 with IL-2 secreting cell line

SUMMARY:
Evaluation of safety and tolerability of four intradermal injections given at two week intervals. In addition the efficacy of transferrinfection was determined by quantifying Interleukin 2 (IL-2), which was locally produced by the implanted, transfected allogenic melanoma cells at the injection sites. Further determination of tumor specific and clinical host responses induced or augmented by the treatment were determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients who fail to respond to conventional therapy or for whom conventional therapy is not available
* Metastatic melanoma (stage IV AJCC) which is surgically or medically incurable because of distant metastatic disease (i.e., a metastasis not in the same lymph node draining area as the primary malignant melanoma). Histologic confirmation of stage IV is required. Measurable disease that can be routinely assessed by physical examination and/or non-invasive radiological procedures
* Karnofsky performance status is at least 60% and life expectancy greater than 4 months
* Male or female, minimum age 18 years
* Written informed consent of the patient in accordance with good clinical practice and local legislation
* Availability of material for autologous Delayed Type Hypersensitivity (DTH) testing (material derived from autologous melanoma metastases and in-house preparation successful) is a requisite for entering the study
* Patients have to undergo biopsy of at least one metastasis before the first and after the last vaccination

Exclusion Criteria:

* Patient who have received any chemotherapy, corticosteroids, radiotherapy (stereotactic irradiation permitted), immunotherapy (e.g. Granulocyte Macrophage Colony Stimulating Factor, Granulocyte Colony Stimulating Factor) or any other investigational drugs in the 4 weeks prior to the first vaccination or prior to surgical removal of tumor specimens for DTH material preparation (patients are not permitted to receive such therapies 4 weeks prior to first cell inoculation except of tumor reductive surgery which are medically indicated)
* Patients with active intracranial metastases (CT/MRI) or choroidal melanoma
* Patients with active autoimmune disease
* Patients with organ allografts
* Patients with evidence of one or more of the following infections: HIV-1, HIV-2, Hepatitis B Virus, Hepatitis C Virus, Human T lymphotropic Virus-1
* Patients with active systemic infections or other major medical illness of the cardiovascular organ system [e.g. coronary heart disease (New York Heart Association class III or IV), history of clinically significant ventricular arrhythmias or angina], coagulation disorder, respiratory or nervous system disorder or with severe endocrinological disease
* Women of childbearing potential with a positive pregnancy test or without appropriate contraception (e.g. IUD [ Intra-Uterine Device], oral contraceptives) until at least 28 days after the last vaccination
* Lactating women
* Impaired renal or hepatic function (serum creatinine > 1.5 mg/dl or creatinine clearance < 75 ml/min). In amendments 1 and 3 serum creatinine levels were changed to 2.5 mg/dl and creatinine clearance was reduced to 30 ml/min
* Impaired hematologic function with:

  * White Blood Count (WBC) < 2500/mm**3 or
  * absolute lymphocyte count < 1500/mm**3 or
  * hemoglobin < 8 g/dl or
  * platelets < 100,000/mm**3
* Evidence for the existence or history of other malignant neoplasms (except adequately treated basal cell carcinoma and carcinoma in situ of the cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 1998-08; Primary Completion 2001-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicity (DLT) | up to 6 weeks
Number of patients with adverse events | up to 28 days after the last vaccination

SECONDARY OUTCOMES:
Grading of local reactions on a 4-point-scale | up to 28 days after the last vaccination
Number of patients with IL-2 transcripts in biopsies of injection sites | 4-6 and 48 hours after first vaccination
Number of patients with delayed type hypersensitivity skin reaction | up to 28 days after the last vaccination
  delayed type hypersensitivity testing
Number of antigen-positive cells in biopsies from metastatic lesions | up to 28 days after the last vaccination
Number of antigen-positive cells in the cellular infiltrate at the vaccination site | up to 28 days after the last vaccination
Number of patients with a positive reaction to Multitest Merieux | up to day 14
  positive reaction: sum of all indurations of all existing reactions => 10 mm (male) or >= 5 mm (female)
Change in T cell proliferation as ratio of post-vaccination to pre-vaccination | up to 28 days after the last vaccination
Change in S-100 beta protein level in serum | up to 28 days after the last vaccination
Number of patients with clinical response | up to 28 days after the last vaccination
  clinical response = complete and partial response
Change in interferon-gamma secretion as ratio of post-vaccination to pre-vaccination | up to 28 days after the last vaccination